CLINICAL TRIAL: NCT03740373
Title: A Phase I, Randomised, Two-Period, Single-Dose, Single-Centre, Crossover Gamma Scintigraphy Study to Assess the Pulmonary Deposition of Technetium-99m Radiolabelled Budesonide, Glycopyrronium and Formoterol Fumarate MDI, Following 3 s and 10 s Breath-Hold, in Healthy Male Subjects
Brief Title: A Study to Assess the Pulmonary Distribution of Budesonide, Glycopyrronium and Formoterol Fumarate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5980C00007
Record Dates: First submitted 2018-08-03; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate; Formoterol Fumarate; Breath Holding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Subjects will receive BGF MDI with 10 s breath hold during Treatment Period 1 and BGF MDI with 3 s breath hold during Treatment Period 2
  Interventions: Drug: BGF MDI (budesonide, glycopyrronium and formoterol fumarate) with 10 s breath hold; Drug: BGF MDI ((budesonide, glycopyrronium and formoterol fumarate) with 3 s breath hold
- Treatment Sequence 2 (Experimental): Subjects will receive BGF MDI with 3 s breath hold during Treatment Period 1 and BGF MDI with 10 s breath hold during Treatment Period 2
  Interventions: Drug: BGF MDI (budesonide, glycopyrronium and formoterol fumarate) with 10 s breath hold; Drug: BGF MDI ((budesonide, glycopyrronium and formoterol fumarate) with 3 s breath hold

INTERVENTIONS:
Drug: BGF MDI (budesonide, glycopyrronium and formoterol fumarate) with 10 s breath hold — Participants will receive a single dose of BGF MDI; the dose will be administered with a 10 s breath-hold.
  Other Names: PT010 with 10 s breath hold
Drug: BGF MDI ((budesonide, glycopyrronium and formoterol fumarate) with 3 s breath hold — Participants will receive a single dose of BGF MDI; the dose will be administered with a 3 s breath-hold.
  Other Names: PT010 with 3 s breath hold

SUMMARY:
This study is a 2 treatment period, single dose crossover, gamma scintigraphy study investigating the deposition in the lungs of a Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler.

This study will be investigating how the drug (known as PT010) is distributed in the lungs following a 10 second or 3 second breath hold.

The study will involve the following visits: 1 screening visits, 2 treatment visits, each separated by around 7 days (each with 1 overnight stay; from the evening before dosing until a minimum of 4 hours post-dose on the morning of Day 1) and a post-study follow up phone call.

The study population will be 10 healthy males, aged between 28 and 50 years of age.

DETAILED DESCRIPTION:
This study is a 2 treatment period, single dose crossover, gamma scintigraphy study investigating the deposition in the lungs of a Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler.

This study will be investigating how the drug (known as PT010) is distributed in the lungs following a 10 second or 3 second breath hold.

This inhaler is intended to be used in the treatment of Chronic Obstructive Pulmonary Disease (COPD), which is a group of diseases which cause lung problems and difficulty breathing.

PT010 contains a combination of 3 marketed drugs called Glycopyrronium, Formoterol Fumarate and Budesonide.

Budesonide is a corticosteroid that works by preventing inflammation and thus can aid in respiratory diseases such as chronic obstructive pulmonary disease. Glycopyrronium & Formoterol Fumarate are bronchodilators which act by relaxing the smooth muscle cells in the trachea and bronchi, allowing greater airflow into the lungs.

To enable us to determine how much of the drug gets into the lungs following different lengths of breath hold, a technique called gamma scintigraphy will be used. Gamma scintigraphy is a technique used to track the movement of a radiolabelled tracer inside the body.

By assessing the amount of PT010 in the lungs following different lengths of breath hold, it is intended that this information will provide guidance as to the most effective way of taking the inhaler.

The study will involve the following visits: 1 screening visits, 2 treatment visits, each separated by around 7 days (each with 1 overnight stay; from the evening before dosing until a minimum of 4 hours post-dose on the morning of Day 1) and a post-study follow up phone call.

The study population will be 10 healthy males, aged between 28 and 50 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 28 and 50 years of age inclusive;
2. Male subject willing to wear a condom and whose partner of child bearing potential uses a highly effective method of contraception (e.g. partner use of intrauterine device (IUD)) or an effective method of contraception, i.e., established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP;
3. Subjects who have a body weight ≥50 kg at the Screening Visit and Subjects with a body mass index (BMI) of 18-30; BMI = body weight (kg) / [height (m)]2.
4. Subject with no clinically significant history of previous allergy / sensitivity to Budesonide, Glycopyrronium and Formoterol Fumarate or any of the excipients contained within the IMP;
5. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 28 days before the first dose of IMP;
6. Subject with a negative urinary drugs of abuse screen, determined within 28 days before the first dose of IMP (N.B. a positive alcohol result may be repeated at Investigator's discretion);
7. Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results;
8. Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before first dose of IMP;
9. Subject with no clinically significant abnormalities in vital signs (e.g., blood pressure/pulse, respiration rate, oral temperature) determined within 28 days before first dose of IMP (Supine BP <140/90 mmHg or resting HR<100 beats per minute);
10. Subject must be available to complete the study (including all follow up contact);
11. Subject must satisfy a medical examiner about their fitness to participate in the study;
12. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subjects with clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, haematological, psychiatric, or other medical illness that would interfere with participation in this study;
2. Subjects with a history of ECG abnormalities including PR>220 msec; QRS complex >120 msec; QT Corrected Using Fridericia's Formula (QTcF) >450 ms; or any significant morphological changes other than non-specific T wave changes;
3. A history of additional risk factors for Torsades de Pointes (e.g., heart failure, family history of Long QT Syndrome);
4. Subjects who have cancer that has not been in complete remission for at least 5 years;
5. Subjects with a FEV1 < 80% of predicted value and/or a FEV1/FVC ratio < 0.7 at screening. Subjects must be able to perform reliable, reproducible pulmonary function test manoeuvres per American Thoracic Society / European Respiratory Society (ATS/ERS) guidelines;
6. Subjects with symptomatic prostatic hypertrophy / prostrate resection within 6 months of screening / bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator;
7. Subjects with a family history of glaucoma or a diagnosis of glaucoma;
8. History of substance-related disorders (with the exception of caffeine-related and nicotine-related disorders) as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM), fourth edition, text revision within 1 year of Screening;
9. History of smoking or the use of nicotine containing products or electronic cigarettes within 3 months of Screening by self-reporting;
10. A positive alcohol or urine drug screen including cotinine for drugs of abuse at the Screening Visit or at the beginning of each treatment period;
11. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMP, unless in the opinion of the Investigator and Sponsor's Responsible Physician the medication will not interfere with the study procedures or compromise subject safety. Paracetamol will be permitted at doses of ≤4 grams/day;
12. Subjects with a history of an allergic reaction or hypersensitivity to the study drugs, or who develop allergic reaction or hypersensitivity to any component of the formulation(s) used in this study including 99mTc;
13. Subjects with a chronic medical condition that requires ongoing treatment with medication;
14. Subjects with a history of major surgery within 4 weeks or minor surgery within 2 weeks of drug administration;
15. Subjects with any flu-like syndrome or other respiratory infections within 2 weeks of drug administration;
16. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study drug non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study related procedures);
17. Subjects with abnormal-glomerular filtration rate (GFR; estimated GFR <90 mL/min/1.73m2) using the Chronic Kidney Disease Epidemiology Collaboration Equation (CKD-EPI);
18. Participation in a study in which radioisotopes were administered within 12 months preceding the first dose of Period 1 of this study, or has been exposed to radiation excess within the last 12 months (e.g., x-rays, handling of radiolabel materials). Radiation excess will be determined on a case-by-case basis following review by the Principal Investigator or designee;
19. Subjects with abnormal findings in a previous chest X ray or CT scan;
20. Subjects who in the opinion of the Investigator are unable to demonstrate acceptable use of the MDI device (including sufficient inspiratory flow rate) and exhalation filter after training;
21. Subjects with any abnormal findings on the 81mKr ventilation scan performed during Treatment Period 1;
22. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction;
23. A clinically significant history of drug or alcohol abuse;
24. Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function);
25. Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).

Ages: 28 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Percentage lung deposition following 10 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The percentage (%) emitted dose of radiolabelled BGF MDI deposited in the lungs following 10 s breath hold.

SECONDARY OUTCOMES:
Percentage lung deposition following 3 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The percentage (%) emitted dose of radiolabelled BGF MDI deposited in the lungs following 3 s breath hold.
Regional airway deposition following 10 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The regional airway deposition ratios including outer to inner (O/I) and central to peripheral (C/P) regions of the radiolabelled BGF MDI following a 10 s breath hold.
Oropharyngeal and stomach deposition following 10 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The fraction of the dose of radiolabelled BGF MDI deposited in the oropharyngeal and stomach regions (expressed as % emitted dose) following a 10 sec breath hold.
Actuator and exhalation filter deposition following 10 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The fraction of the dose of radiolabelled BGF MDI deposited on the actuator (expressed as % ex-valve dose) and exhalation filter (expressed as % emitted dose) following a 10 s breath hold.
Regional airway deposition following 3 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The regional airway deposition ratios including outer to inner (O/I) and central to peripheral (C/P) regions of the radiolabelled BGF MDI following a 3 s breath hold.
Oropharyngeal and stomach deposition following 3 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The fraction of the dose of radiolabelled BGF MDI deposited in the oropharyngeal and stomach regions (expressed as % emitted dose) following a 3 s breath hold.
Actuator and exhalation filter deposition following 3 s breath hold | Day 1 (of either Treatment Period 1 or 2)
  The fraction of the dose of radiolabelled BGF MDI deposited on the actuator (expressed as % ex-valve dose) and exhalation filter (expressed as % emitted dose) following a 3 s breath hold.

OTHER OUTCOMES:
Number of TEAEs | Day 1 to Follow-up (Day 7-14 post-dose)
  Number of TEAEs
Number of subjects reporting at least 1 Treatment Emergent Adverse Event | Day 1 to Follow-up (Day 7-14 post-dose)
  Number of subjects reporting at least 1 Treatment Emergent Adverse Event
Number of subjects reporting at least 1 serious Treatment Emergent Adverse Event | Day 1 to follow-up (Day 7-14 post dose)
  Number of subjects reporting at least 1 serious Treatment Emergent Adverse Event
Number of subjects reporting at least 1 Treatment Emergent Adverse Event leading to withdrawal from the study | Day 1 to Follow-up (Day 7-14 post dose)
  Number of subjects reporting at least 1 Treatment Emergent Adverse Event leading to withdrawal from the study
Number of subjects reporting Treatment Emergent Adverse Events by severity and relationship to IMP. | Day 1 to Follow-up (Day 7-14 post-dose)
  Number of subjects reporting Treatment Emergent Adverse Events by severity and relationship to IMP.
Percentage of subjects reporting at least 1 Treatment Emergent Adverse Event | Day 1 to Follow-up (Day 7-14 post-dose)
  Percentage of subjects reporting at least 1 Treatment Emergent Adverse Event
Percentage of subjects reporting at least 1 serious Treatment Emergent Adverse Event | Day 1 to follow-up (Day 7-14 post dose)
  Percentage of subjects reporting at least 1 serious Treatment Emergent Adverse Event
Percentage of subjects reporting at least 1 Treatment Emergent Adverse Event leading to withdrawal from the study | Day 1 to Follow-up (Day 7-14 post dose)
  Percentage of subjects reporting at least 1 Treatment Emergent Adverse Event leading to withdrawal from the study
Percentage of subjects reporting Treatment Emergent Adverse Events by severity and relationship to IMP. | Day 1 to Follow-up (Day 7-14 post-dose)
  Percentage of subjects reporting Treatment Emergent Adverse Events by severity and relationship to IMP.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Israel, Principal Investigator — Simbec Research
Locations (1):
- Research Site, Pentrebach, United Kingdom